CLINICAL TRIAL: NCT04508556
Title: Performance Assessment of SARS-CoV-2 Detection Through Analysis of Exhaled Breath Aerosols
Brief Title: Performance Assessment of SARS-CoV-2 Detection Breath Biopsy - SARS-CoV-2 Study
Acronym: COVID
Status: Completed | Type: Observational
Sponsor: Owlstone Ltd (Industry)
Collaborators: OLVG (Network); Maastricht University (Other)
Responsible Party: Sponsor
Other Study IDs: SARS-CoV-2 study
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — The face mask will be placed onto the subject's face, covering his/her nose and mouth, head straps will be used to ensure that the face mask is kept in place for the duration of the test. This mask will contain a material designed to capture exhaled respiratory droplets and/or aerosols. Several iterations of these impaction and filtration devices may be used to optimize functional attributes of the material for capture of COVID. These materials will always have a proven safety for use with humans.
  Subjects can talk, cough and sneeze in the mask or can temporarily remove the mask if uncomfortable, to drink some water etc if required. Total collection time spread across two masks will not exceed one hour
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Device: Breath Biopsy face masks with removable filters and fitted PVA strip — Device developed for collection of breath samples
Diagnostic Test: Nasopharyngeal swab — Is a method for collecting a clinical test sample of nasal secretions from the back of the nose and throat.
Diagnostic Test: oropharyngeal swabs — Is a method for collecting a clinical test sample from the back of the throat.

SUMMARY:
The primary aim of this study is to investigate the performance of Breath Biopsy RD for the detection of SARS-CoV-2 in both a clinical and at home setting.

DETAILED DESCRIPTION:
This study aims to evaluate Owlstone Medical's Breath Biopsy RD Collectors for the detection of SARS-CoV-2 infection. These single use disposable breath capture devices can be used independently by individuals and shipped to be analysed in a central lab for the presence of SARS-CoV-2 using established existing PCR assays available in any reference lab. The aerosol collectors furthermore directly sample exhaled breath aerosols. As such they directly sample the primary transmission route for the virus. This could result in a higher rate of retrieval of viral RNA in infected individuals thereby increasing the sensitivity of the applied PCR assay. This is underpinned by the fact that CT abnormalities in the lower airways appear to occur prior to upper respiratory tract samples becoming positive in cases suffering from nCOVID19, suggesting lower airway viral loads could be higher. Combined, this could enable more widespread access to diagnostics, reduce the need for repeat testing, decrease the need for healthcare professionals to perform diagnostic tests and reduce cross-contamination risk.

ELIGIBILITY:
Inclusion Criteria:

* Any adult >18 years with either a confirmed (phase 1) or suspected (phase 2&3) SARS-CoV-2 infection will be eligible to participate in this study.

Exclusion Criteria:

* Subject who are deemed unlikely to be able to maintain oxygen saturation of greater than 90% while breathing room air for 30 seconds
* Subject who require non-invasive ventilation or high flow nasal oxygen
* Subject who require inotropic medication to maintain adequate organ perfusion
* Subject who have a communication barrier and / or unable to comply with the instructions to use the Breath Biopsy test

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The inclusion and exclusion criteria for the various study populations are detailed above. General inclusion and exclusion criteria which apply to all study subjects are detailed followed by indication specific criteria are also detailed for both inclusion and exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2020-12-19 (Actual); Study Completion 2020-12-19 (Actual)

PRIMARY OUTCOMES:
Positive control for technical validation | 1 year
  The purpose of this stage is to confirm the optimal extraction protocol to detect the presence of SARS-CoV-2 from the aerosols captured in the Breath Biopsy RD device. Up to two Breath Biopsy RD sample will be collected alongside a nasopharyngeal. The swab obtained during this stage is to be analysed in parallel to the extracted breath aerosols in the lab of the lab and will be used as a positive control.

SECONDARY OUTCOMES:
Evaluation of test performance | 1 year
  The aim is to assess the test performance of the Breath Biopsy RD devices in a real live clinical setting. Subjects with a high clinical suspicion of nCOVID-19 based on clinical triage will be requested to participate. A single Breath Biopsy RD collector will be collected in parallel with the standard diagnostic work-up consisting of a CT-scan and a nasopharyngeal swab.

OTHER OUTCOMES:
Evaluation of at home test | 1 year
  The aim of the final outcome is to evaluate the performance and acceptability of using the Breath Biopsy RD as an at home test for identification of the presence of SARS-CoV-2. The OLVG phone application used for triage of the presence of nCOVID-19 will be used to identify subjects at the highest risk of having nCOVID-19. These subjects will be sent a Breath Biopsy RD collector and oropharyngeal swab for at home testing. Any subject who has a positive Breath Biopsy test for SARS-CoV-2 will be contacted and advised to receive a nasopharyngeal test for assessment of viral presence. Both tests will be self-administered to mimic an at home use scenario. The performance of both tests will be confirmed from the perspective of 1. Adherence 2. Subject comfort 3. Number of SARS-CoV-2 positive cases.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Savelkoul,, Study Chair — OLVG; Paul Bresser, Study Chair — Maastricht
Locations (1):
- OLVG, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No